CLINICAL TRIAL: NCT07017127
Title: Remission of Type 2 Diabetes With Mediterranean Diet, Physical Activity and Psychological Support: a Randomized Clinical Trial
Brief Title: Remission of Type 2 Diabetes With Lifestyle Intervention
Acronym: REMeDI2ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Ivana Kolcic, Professor, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRZZ-IP-2024-05-3757; 2181-198-03-04-24-0117 (Other: University of Split School of Medicine, Croatia); 2181-147/01-06/LJ.Z.-24-02 (Other: Clinical Hospital Centre Split, Croatia); 2181-149-18-24-002 (Other: Split-Dalmatia Health Center, Croatia)
Record Dates: First submitted 2025-03-08; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus Type 2; Obese Diabetics
Keywords: diabetes remission; Mediterranean diet; physical activity; stress; weight loss; healthy lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Weight Loss | interventions — Diet, Mediterranean; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle intervention group (Experimental): The intervention will consist of the following elements:
  1. Mediterranean diet - personalized nutritional recommendation based on the modern pyramid of the Mediterranean diet (44), additionally adjusted based on the current nutritional status of the subjects (tested through anthropometric and body composition parameters), and considering the level of physical activity during free time and professional requirements
  2. Physical activity - emphasis on reducing sedentary behavior and including a daily regime of aerobic exercises, and exercises for muscle strength and endurance 2 times a week
  3. Psychological support and intervention - group and individual counselling of subjects on effective ways of coping with stress
  4. Positive and supportive interpersonal relationships - implementation of the intervention in small groups, which will be formed primarily as support groups (12 subjects per group) - weekly meetings, counselling and workshops, group exercise (walking)
  Interventions: Behavioral: Mediterranean diet; Behavioral: Physical activity intervention; Behavioral: Psychological intervention
- Control group (No Intervention): Subjects in the control group will receive a short brochure that will be created for the purposes of this project on the importance of healthy lifestyle habits in people diagnosed with DM2, as well as advice and recommendations from a specialists for practicing healthy eating and physical activity. Furthermore, the subjects of the control group will receive regular clinical care within the framework of the health care system. At the same time intervals as the subjects of the experimental group, these subjects will be invited for a clinical examination, carrying out all measurements and tests, filling out questionnaires and providing biological samples (fasting blood and urine).

INTERVENTIONS:
Behavioral: Mediterranean diet — Exclusion of highly processed food products and beverages, introduction of a diet according to the modern pyramid of the Mediterranean diet (44). Subjects will be recommended to reduce as much as possible the use of plastic food and drinks containers. The nutritionist will create personalized nutritional recommendation, with a moderate reduction in caloric intake (quantified by calculating the basal metabolism and ideal body mass of each subject, and the whole day's energy consumption). The goal of this part of the intervention is to achieve a weight loss of at least 0.5 kg every week, by reducing caloric intake by 300-500 kcal. The nutritionist will create sample menus throughout the day, for 30 days, to make it easier for subjects to follow this part of the intervention. In addition, each subject of the experimental group will receive a total of six liters of extra virgin olive oil (one liter per month for 6 months).
  Arms: Lifestyle intervention group
Behavioral: Physical activity intervention — Participants will be involved in aerobic activities expertly guided by kinesiologist (Nordic walking) every day for 45-60 minutes, spent in nature or indoors in case of unfavorable weather. Along with Nordic walking, participants will be involved in organized muscle strength and endurance exercises twice a week for 60 minutes with the use of external loads (elastic bands, small weights), and mobility, balance and coordination will also be developed. All training programs will be conducted by trained kinesiologists who will instruct, monitor and correct participants in order to perform the exercises correctly and get the maximum effect on the targeted motor skills. Nordic walking, resistance exercise, and a combination of aerobic activity and resistance exercise have been shown to be effective in improving cardiometabolic parameters, physical fitness, and quality of life in people with DM2.
  Arms: Lifestyle intervention group
Behavioral: Psychological intervention — Support group meetings discussing mental health topics and encouraging change through the adoption of healthy lifestyle habits. Psycho-educational component, stimulating group environment for sharing personal experiences, motivation and becoming aware of emotions and resistance. The specific topics of individual group meetings will be: stress and stress management, relaxation techniques (breathing techniques, autogenic training, progressive muscle relaxation techniques and guided fantasies), emotion management (recognition of negative beliefs and thought patterns, awareness and management of emotional reactions), interpersonal skills in the function of self-care (awareness and communication of one's own needs through assertive communication techniques), self-care through the adoption of healthy habits (motivation, adoption of habits and planning), conscious eating and the alike, creating a list of SMART goals (45).
  Arms: Lifestyle intervention group

SUMMARY:
The goal of this clinical trial is to achieve diabetes type 2 (DM2) remission using intensive lifestyle intervention.

The main questions it aims to answer are:

* Does intensive lifestyle intervention (including Mediterranean diet with a caloric deficit, daily physical activity, increase in stress resilience and group support) lead to DM2 remission (HbA1c<6.5%, without medications)
* Can intensive lifestyle intervention (including Mediterranean diet with a caloric deficit, daily physical activity, increase in stress resilience and group support) result to weight loss of >15 kg
* Does intensive lifestyle intervention result in any side effects (secondary outcome)

Researchers will compare intensive lifestyle intervention to the usual clinical care (control group).

Participants in the experimental group will:

* eat Mediterranean diet with a caloric deficit
* perform daily physical activity
* increase their stress resilience with psychosocial support of the group
* enroll weekly in individual and group counseling and workshops for 6 months, following with 1.5 years of follow-up

DETAILED DESCRIPTION:
Type 2 diabetes (diabetes mellitus type 2, DM2) is a leading clinical and public health problem, with a global prevalence that is rapidly increasing and reaching pandemic proportions. According to the International Diabetes Federation (IDF), 537 million adults between the ages of 20 and 79 in the world have type 2 diabetes (DM2), and it is predicted that this number will increase to 643 million by 2030 and 783 million by 2045. According to the data of the National Register of Persons with DM2 (CroDiab) 337,774 persons with DM2 type 2 were registered in Croatia in 2022.

DM2 increases the risk for cardiovascular diseases, blindness, kidney failure and amputation of the lower limbs, thereby significantly affecting the quality of life of the patients. Additionally, it is well known that people with DM2 often have obstructive sleep apnea (OSA). Therefore, active screening for an OSA diagnosis and its treatment in patients with DM2 is extremely important for the prognosis and successful treatment of DM2, especially since it has been shown that CPAP treatment, along with body weight reduction, is associated with a reduction in HbA1c in morbidly obese patients with severe OSA.

The increased prevalence of DM2 is inextricably linked to the change in lifestyle and the transition to a "western" lifestyle, which implies an abundance of energy-rich foods and reduced physical activity, with a subsequent increase in obesity. Looking at individual components of the diet, it has been shown that sweetened beverages, refined grains and processed meat increase the risk of developing DM2. On the other hand, green leafy vegetables, dairy products, whole grains, nuts, legumes, moderate amounts of alcohol and coffee are associated with a reduction in this risk. Considering not only the individual nutrients in the diet but the entire nutrition pattern, the Mediterranean diet stands out with its numerous protective effects on the health of the organism. Epidemiological and interventional studies have shown the protective effect of the Mediterranean diet in chronic inflammation, insulin resistance, and metabolic syndrome. The Mediterranean diet is best known for its protective cardiovascular effect, which has been shown in a number of studies, meta-analyses and systematic reviews. Among other things, this type of diet supports healthy aging (reaching the age of 70 and over without chronic diseases, such as DM2, kidney disease, respiratory diseases, cancer or Parkinson's disease, and without significant decline in mental and cognitive function).

Losing excess body weight is a key factor in achieving remission of DM2, therefore it is important to look at the evidence of how different dietary patterns can promote weight loss. Comparing low-carbohydrate, low-fat, and Mediterranean diet showed that both the Mediterranean diet and the low-carbohydrate diet were superior in achieving weight loss compared to the low-fat diet. Moreover, these two dietary patterns also showed significant metabolic benefits, such as reduced CRP, reduced fasting glucose and increased insulin sensitivity. In the PREDIMED study, it was shown that a Mediterranean diet supplemented with nuts or extra virgin olive oil reduces the risk of death from stroke by 30%. In addition, there was a significant reduction in the incidence of DM2 in subjects on the Mediterranean diet, independent of weight loss or the subjects' physical activity. Hence, besides weight loss, the quality of nutrition is a valuable factor in the prevention of DM2. The Mediterranean diet is based primarily on unprocessed food of plant origin (vegetables, fruits, legumes, whole grains, nuts). Moderate consumption of fish, seafood and dairy products is encouraged, as well as avoiding red and processed meat. The main source of fat in the Mediterranean diet is extra virgin olive oil. Apart from water as the main drink, wine can be enjoyed in moderation with a meal.

DM2 is considered to be an incurable, chronic and progressive disease. However, several studies recently showed that it is possible to achieve a remission of the disease. It is considered that the remission of DM2 has been achieved if Hba1c is less than 6.5%, without the use of blood glucose-lowering drugs for at least 3 months. Body weight control is the most important aspect of DM2 treatment, with weight reduction leading to reduced morbidity and mortality in these patients. The results of several studies have shown that weight loss of at least 10-15 kg leads to normalization of blood glucose levels in people who were relatively recently diagnosed with DM2. The DIRECT study showed that an intensive and structured weight management program delivered in primary care can result in significant weight loss and diabetes remission among adults with newly diagnosed diabetes. Remission of DM2 was achieved in 46% of subjects who lost an average of 10 kg, after one year. After two years, 36% of subjects were still in remission, with an average of 8 kg lost.

Another study achieved excellent DM2 remission results using dietary modification. The Diabetes Intervention Accentuating Diet and Enhancing Metabolism (DIADEM-I) study followed the effect of a 12-month intensive lifestyle intervention, which consisted of complete meal replacement, in subjects who were younger than 50 years and had been diagnosed with DM2 in the previous 3 years. DM2 remission was achieved in 61% of subjects who lost 15% of their initial weight.

Procedures:

Two groups of subjects will be included in the study: an experimental group and a control group, using the same criteria for the inclusion and exclusion.

Experimental group: the intervention will consist of the following elements:

1. Mediterranean diet - personalized nutritional recommendation based on the modern pyramid of the Mediterranean diet, additionally adjusted based on the current nutritional status of the subjects (tested through anthropometric and body composition parameters), and considering the level of physical activity during free time and professional requirements
2. Physical activity - emphasis on reducing sedentary behavior and including a daily regime of aerobic exercises, and exercises for muscle strength and endurance 2 times a week
3. Psychological support and intervention - group and individual counselling of subjects on effective ways of coping with stress
4. Positive and supportive interpersonal relationships - implementation of the intervention in small groups, which will be formed primarily as support groups (12 subjects per group) - weekly meetings, counselling and workshops, group exercise (walking), during which education and counselling on nutrition, physical activity and psychological determinants of health will take place.

Detailed description of the intervention, consisting of changes in lifestyle habits in four domains:

The nutritional intervention will consist of the exclusion of highly processed food products and beverages containing free simple sugars, along with the introduction of a diet according to the modern pyramid of the Mediterranean diet. In addition, subjects will be recommended to reduce (and when possible, to exclude) the use of plastic drinking containers, plastic containers for food preparation and storage, in order to reduce exposure to endocrine disruptors. For each subject, the nutritionist will create a personalized nutritional recommendation, with a moderate reduction in caloric intake, in order to ensure a gradual loss of body weight. The required level of caloric reduction will be quantified by calculating the basal metabolism and ideal body mass of each subject of the experimental group (based on anthropometric measurement and determination of body composition), and the whole day's energy consumption will be determined, considering the physical activity of the person and energy necessary for digestion and assimilation of nutrients. The goal of this part of the intervention is to achieve a weight loss of at least 0.5 kg every week, or approximately 2 kg per month, which will be achieved by reducing caloric intake by 300-500 kcal. Personal preferences of the subjects towards certain foods will be considered, all in accordance with the Mediterranean diet pyramid. The nutritionist will create sample menus throughout the day, for 30 days, to make it easier for subjects to follow this part of the intervention. In addition, each subject of the experimental group will receive a total of six liters of extra virgin olive oil (one liter per month, during the six months of the intervention), considering that olive oil is an indispensable element of the Mediterranean diet, in order to avoid financial burden on the subjects. Investigators expect this will increase the subjects' compliance.

Physical activity intervention: Participants will be involved in aerobic activities expertly guided by kinesiologist (Nordic walking) every day for 45-60 minutes, spent in nature or indoors in case of unfavorable weather. Along with Nordic walking, participants will be involved in organized muscle strength and endurance exercises twice a week for 60 minutes with the use of external loads (elastic bands, small weights), and mobility, balance and coordination will also be developed. All training programs will be conducted by trained kinesiologists who will instruct, monitor and correct participants in order to perform the exercises correctly and get the maximum effect on the targeted motor skills. Nordic walking, resistance exercise, and a combination of aerobic activity and resistance exercise have been shown to be effective in improving cardiometabolic parameters, physical fitness, and quality of life in people with DM2.

Psychological intervention will consist of support groups, where of mental health topics and encouraging change through the adoption of healthy lifestyle habits will be discussed. In addition to the psycho-educational component, participants in the stimulating group environment will have the opportunity to share personal experiences, motivation and become aware of emotions and resistance, which is crucial in achieving and maintaining change. The specific topics of individual group meetings will be: stress and stress management, relaxation techniques (breathing techniques, autogenic training, progressive muscle relaxation techniques and guided fantasies), emotion management (recognition of negative beliefs and thought patterns, awareness and management of emotional reactions), interpersonal skills in the function of self-care (awareness and communication of one's own needs through assertive communication techniques), self-care through the adoption of healthy habits (motivation, adoption of habits and planning), conscious eating and the alike. Each subject will create for himself a list of SMART goals that she/he wants to achieve during his participation in the project (Specific, Measurable, Achievable, Relevant, and Time-Bound).

Positive and supportive interpersonal relationships can result in more sustainable effects on behaviors change in patients with chronic non-communicable diseases, and are an important component of chronic disease self-management, and can be an effective resource in patients trying to lose excess weight.

Control group: subjects of the control group will receive a short brochure that will be created for the purposes of this project on the importance of healthy lifestyle habits in people diagnosed with DM2, as well as advice and recommendations from a specialist for practicing healthy eating and physical activity. Furthermore, the subjects of the control group will receive regular clinical care within the framework of the health care system. At the same time intervals as the subjects of the experimental group, these subjects will be invited for a clinical examination, carrying out all measurements and tests, filling out questionnaires and providing biological samples (fasting blood and urine).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes diagnosis
* incident cases or diagnosed not more than 7 years ago
* body mass index of 27-45 kg/m²

Exclusion Criteria:

* mobility restriction
* use of mobility aids
* insulin therapy
* HbA1c >12%
* TSH >10 mU/L
* heart failure (NYHA III, NYHA IV)
* use of obesity pharmacotherapy (orlistat, GLP-1 receptor agonists, GLP-1/GIP dual agonists) for less than 6 months
* weight loss greater than 5 kg in the last 6 months
* chronic kidney disease and estimated glomerular filtration rate <30 ml/min/1.73 m2
* active treatment of proliferative diabetic retinopathy with anti-VEGF
* heart attack or stroke in the past 1 year
* active malignant disease diagnosed in the past 1 year
* eating disorders
* pregnancy or pregnancy planning
* substance abuse
* learning disabilities
* acute episode of severe depression
* current use of antipsychotics
* food allergy

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Remission of diabetes mellitus type 2 | 24 months
  Change of HbA1c to <6.5%, without the use of blood glucose lowering therapy for the past 3 months

SECONDARY OUTCOMES:
Weight loss | 24 months
  Loss of body weight of ≥15 kg
Adverse events | 24 months
  Any adverse event associated with each of the interventions (nutritional, physical activity, psychological)

OTHER OUTCOMES:
Additional benefits | 24 months
  change in arterial function measured as pulse wave velocity (PWV)
Additional benefits | 24 months
  change in Advanced Glycation End Products measured using AGE Reader mu (DiagnOptics)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Kolčić, Prof, MD, PhD, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esposito K, Maiorino MI, Petrizzo M, Bellastella G, Giugliano D. The effects of a Mediterranean diet on the need for diabetes drugs and remission of newly diagnosed type 2 diabetes: follow-up of a randomized trial. Diabetes Care. 2014 Jul;37(7):1824-30. doi: 10.2337/dc13-2899. Epub 2014 Apr 10. PMID 24722497
- [Background] Gutierrez-Mariscal FM, Alcala-Diaz JF, Quintana-Navarro GM, de la Cruz-Ares S, Torres-Pena JD, Cardelo MP, Arenas-Larriva AP, Malagon MM, Romero-Cabrera JL, Ordovas JM, Perez-Martinez P, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Changes in quantity plant-based protein intake on type 2 diabetes remission in coronary heart disease patients: from the CORDIOPREV study. Eur J Nutr. 2023 Jun;62(4):1903-1913. doi: 10.1007/s00394-022-03080-x. Epub 2023 Mar 4. PMID 36869909
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Kelly T, Irvine K, Peters C, Zhyzhneuskaya S, Hollingsworth KG, Adamson AJ, Sniehotta FF, Mathers JC, McIlvenna Y, Welsh P, McConnachie A, McIntosh A, Sattar N, Taylor R. 5-year follow-up of the randomised Diabetes Remission Clinical Trial (DiRECT) of continued support for weight loss maintenance in the UK: an extension study. Lancet Diabetes Endocrinol. 2024 Apr;12(4):233-246. doi: 10.1016/S2213-8587(23)00385-6. Epub 2024 Feb 26. PMID 38423026
- [Background] Taheri S, Zaghloul H, Chagoury O, Elhadad S, Ahmed SH, El Khatib N, Amona RA, El Nahas K, Suleiman N, Alnaama A, Al-Hamaq A, Charlson M, Wells MT, Al-Abdulla S, Abou-Samra AB. Effect of intensive lifestyle intervention on bodyweight and glycaemia in early type 2 diabetes (DIADEM-I): an open-label, parallel-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2020 Jun;8(6):477-489. doi: 10.1016/S2213-8587(20)30117-0. PMID 32445735
- [Background] Chimoriya R, Mitlehner K, Khoo CL, Osuagwu UL, Thomson R, Si L, Lean M, Simmons D, Piya MK. Translation of a Diabetes Remission Service into Australian Primary Care: Findings from the Evaluation of DiRECT-Australia. J Diabetes Res. 2024 Feb 8;2024:2350551. doi: 10.1155/2024/2350551. eCollection 2024. PMID 38361965
- [Background] Al-Mrabeh A, Hollingsworth KG, Shaw JAM, McConnachie A, Sattar N, Lean MEJ, Taylor R. 2-year remission of type 2 diabetes and pancreas morphology: a post-hoc analysis of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2020 Dec;8(12):939-948. doi: 10.1016/S2213-8587(20)30303-X. Epub 2020 Oct 5. PMID 33031736
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132
- [Background] Dixon JB, O'Brien PE, Playfair J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA. 2008 Jan 23;299(3):316-23. doi: 10.1001/jama.299.3.316. PMID 18212316
- [Background] Sjostrom L. Review of the key results from the Swedish Obese Subjects (SOS) trial - a prospective controlled intervention study of bariatric surgery. J Intern Med. 2013 Mar;273(3):219-34. doi: 10.1111/joim.12012. Epub 2013 Feb 8. PMID 23163728
- [Background] Sjostrom L, Peltonen M, Jacobson P, Ahlin S, Andersson-Assarsson J, Anveden A, Bouchard C, Carlsson B, Karason K, Lonroth H, Naslund I, Sjostrom E, Taube M, Wedel H, Svensson PA, Sjoholm K, Carlsson LM. Association of bariatric surgery with long-term remission of type 2 diabetes and with microvascular and macrovascular complications. JAMA. 2014 Jun 11;311(22):2297-304. doi: 10.1001/jama.2014.5988. PMID 24915261
- [Background] Henry RR, Scheaffer L, Olefsky JM. Glycemic effects of intensive caloric restriction and isocaloric refeeding in noninsulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1985 Nov;61(5):917-25. doi: 10.1210/jcem-61-5-917. PMID 4044780
- [Background] Riddle MC, Cefalu WT, Evans PH, Gerstein HC, Nauck MA, Oh WK, Rothberg AE, le Roux CW, Rubino F, Schauer P, Taylor R, Twenefour D. Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes. Diabetes Care. 2021 Aug 30;44(10):2438-44. doi: 10.2337/dci21-0034. Online ahead of print. PMID 34462270
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Samieri C, Sun Q, Townsend MK, Chiuve SE, Okereke OI, Willett WC, Stampfer M, Grodstein F. The association between dietary patterns at midlife and health in aging: an observational study. Ann Intern Med. 2013 Nov 5;159(9):584-91. doi: 10.7326/0003-4819-159-9-201311050-00004. PMID 24189593
- [Background] Rosato V, Temple NJ, La Vecchia C, Castellan G, Tavani A, Guercio V. Mediterranean diet and cardiovascular disease: a systematic review and meta-analysis of observational studies. Eur J Nutr. 2019 Feb;58(1):173-191. doi: 10.1007/s00394-017-1582-0. Epub 2017 Nov 25. PMID 29177567
- [Background] Tang C, Wang X, Qin LQ, Dong JY. Mediterranean Diet and Mortality in People with Cardiovascular Disease: A Meta-Analysis of Prospective Cohort Studies. Nutrients. 2021 Jul 29;13(8):2623. doi: 10.3390/nu13082623. PMID 34444786
- [Background] Esposito K, Marfella R, Ciotola M, Di Palo C, Giugliano F, Giugliano G, D'Armiento M, D'Andrea F, Giugliano D. Effect of a mediterranean-style diet on endothelial dysfunction and markers of vascular inflammation in the metabolic syndrome: a randomized trial. JAMA. 2004 Sep 22;292(12):1440-6. doi: 10.1001/jama.292.12.1440. PMID 15383514
- [Background] Esposito K, Giugliano D. Diet and inflammation: a link to metabolic and cardiovascular diseases. Eur Heart J. 2006 Jan;27(1):15-20. doi: 10.1093/eurheartj/ehi605. Epub 2005 Oct 11. PMID 16219650
- [Background] Ley SH, Hamdy O, Mohan V, Hu FB. Prevention and management of type 2 diabetes: dietary components and nutritional strategies. Lancet. 2014 Jun 7;383(9933):1999-2007. doi: 10.1016/S0140-6736(14)60613-9. PMID 24910231
- [Background] Uusitupa M, Khan TA, Viguiliouk E, Kahleova H, Rivellese AA, Hermansen K, Pfeiffer A, Thanopoulou A, Salas-Salvado J, Schwab U, Sievenpiper JL. Prevention of Type 2 Diabetes by Lifestyle Changes: A Systematic Review and Meta-Analysis. Nutrients. 2019 Nov 1;11(11):2611. doi: 10.3390/nu11112611. PMID 31683759
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] de Pablos-Velasco P, Parhofer KG, Bradley C, Eschwege E, Gonder-Frederick L, Maheux P, Wood I, Simon D. Current level of glycaemic control and its associated factors in patients with type 2 diabetes across Europe: data from the PANORAMA study. Clin Endocrinol (Oxf). 2014 Jan;80(1):47-56. doi: 10.1111/cen.12119. Epub 2013 May 6. PMID 23194193
- [Background] Colditz GA, Willett WC, Rotnitzky A, Manson JE. Weight gain as a risk factor for clinical diabetes mellitus in women. Ann Intern Med. 1995 Apr 1;122(7):481-6. doi: 10.7326/0003-4819-122-7-199504010-00001. PMID 7872581
- [Background] Tasbakan MS, Grote L, Hedner J, Kvamme JA, Verbraecken J, McNicholas WT, Roisman G, Tkacova R, Bonsignore MR, Saaresranta T, Steiropoulos P, Marrone O, Basoglu OK; ESADA Collaborators. Positive airway pressure (PAP) treatment reduces glycated hemoglobin (HbA1c) levels in obstructive sleep apnea patients with concomitant weight loss: Longitudinal data from the ESADA. J Sleep Res. 2021 Oct;30(5):e13331. doi: 10.1111/jsr.13331. Epub 2021 May 14. PMID 33987873
- [Background] Al-Saeed AH, Constantino MI, Molyneaux L, D'Souza M, Limacher-Gisler F, Luo C, Wu T, Twigg SM, Yue DK, Wong J. An Inverse Relationship Between Age of Type 2 Diabetes Onset and Complication Risk and Mortality: The Impact of Youth-Onset Type 2 Diabetes. Diabetes Care. 2016 May;39(5):823-9. doi: 10.2337/dc15-0991. Epub 2016 Mar 22. PMID 27006511
- [Background] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Background] Hillier TA, Pedula KL. Characteristics of an adult population with newly diagnosed type 2 diabetes: the relation of obesity and age of onset. Diabetes Care. 2001 Sep;24(9):1522-7. doi: 10.2337/diacare.24.9.1522. PMID 11522693
- [Background] Abelleira R, Zamarron C, Riveiro V, Casal A, Toubes ME, Rabade C, Ricoy J, Lama A, Rodriguez-Nunez N, Ferreiro L, Rodriguez-Ozores J, Valdes L. Relationship between obstructive sleep apnea and type 2 diabetes mellitus. Med Clin (Barc). 2024 Apr 26;162(8):363-369. doi: 10.1016/j.medcli.2023.11.014. Epub 2024 Jan 13. English, Spanish. PMID 38220552
- [Background] Storgaard H, Mortensen B, Almdal T, Laub M, Tarnow L. At least one in three people with Type 2 diabetes mellitus referred to a diabetes centre has symptomatic obstructive sleep apnoea. Diabet Med. 2014 Nov;31(11):1460-7. doi: 10.1111/dme.12477. Epub 2014 May 20. PMID 24766227